CLINICAL TRIAL: NCT03594227
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of ATI-501 Oral Suspension Compared to Placebo in Adult Subjects With Alopecia Areata, Alopecia Universalis or Alopecia Totalis
Brief Title: ATI-501 Oral Suspension Compared to Placebo in Subjects With Alopecia Areata, Alopecia Universalis or Alopecia Totalis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ATI-501-AUAT-201
Record Dates: First submitted 2018-06-26; First posted 2018-07-20 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-06

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — BID protein, human; Administration, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 400mg BID (Low dose) (Active Comparator): ATI-501 low dose - oral administration
  Interventions: Drug: ATI-501 400mg BID (Low dose)
- 600mg BID (Mid dose) (Active Comparator): ATI-501 mid dose - oral administration
  Interventions: Drug: ATI-501 600mg BID (Mid dose)
- 800mg BID (High dose) (Active Comparator): ATI-501 high dose - oral administration
  Interventions: Drug: ATI-501 800mg BID (High dose)
- Placebo (Placebo Comparator): Placebo - oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATI-501 400mg BID (Low dose) — ATI-501 400mg BID oral low dose for oral administration
  Other Names: Active comparator: Low dose
  Arms: 400mg BID (Low dose)
Drug: ATI-501 600mg BID (Mid dose) — ATI-501 600mg BID oral mid dose for oral administration
  Other Names: Comparator : Mid dose
  Arms: 600mg BID (Mid dose)
Drug: ATI-501 800mg BID (High dose) — ATI-501 800mg BID high dose for oral administration
  Other Names: Comparator: high dose - oral administration
  Arms: 800mg BID (High dose)
Drug: Placebo — Placebo - oral administration
  Arms: Placebo

SUMMARY:
This Phase 2, multicenter, randomized study will evaluate the safety, tolerability and efficacy of ATI-501 for the treatment of Alopecia Areata (AA), Alopecia Universalis (AU) or Alopecia Totalis (AT) in adult subjects.

DETAILED DESCRIPTION:
This Phase 2, multicenter, randomized study will evaluate the safety, tolerability and efficacy of ATI-501 for the treatment of Alopecia Areata (AA), Alopecia Universalis (AU) or Alopecia Totalis (AT) in adult subjects. Subjects will be required to have a clinical diagnosis of stable AA, AU, or AT. A total of approximately 80 subjects will be randomized.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for participation in the study:

1. Able to comprehend and willing to sign an Informed Consent Form (ICF).
2. Male or non-pregnant, non-nursing female ≥ 18 years old at the time of informed consent.
3. Have a clinical diagnosis of stable Alopecia Areata (AA), Alopecia Universalis (AU), or Alopecia Totalis (AT).
4. If the subject is a woman of childbearing potential (WOCBP), she must have:

   * Negative urine and serum pregnancy tests at Screening (Visit 1); and
   * A negative urine pregnancy test at Baseline (Visit 2); and
   * Agree to not be planning a pregnancy during the study duration and use a highly effective method of contraception for the duration of the study and 30 days after the last dose of study medication. (Refer to Section 8.4.2).
5. Be in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the subject or which might expose the subject to an unacceptable risk by study participation.
6. Be willing to maintain the same hair style and hair dyeing throughout the study period.
7. Subjects taking hormonal replacement therapies must be on stable doses for 6 months prior to enrollment and remain on a maintenance dose throughout the study.
8. Subjects taking thyroid replacement medication must be on stable doses for 6 months prior to enrollment and remain on a maintenance dose throughout the study.
9. Sexually active male subjects whose partner is a WOCBP must agree to use a barrier method of contraception from the first dose of study medication to at least 30 days after the last dose of study medication.

Exclusion Criteria:

Subjects are excluded from this study if any 1 or more of the following criteria is met:

1. Females who are nursing, pregnant, or planning to become pregnant for the duration of the study and up to 30 days after the last dose of study medication.
2. Diffuse AA or a history of an atypical pattern of AA.
3. Concomitant hair loss disorder (by history or physical exam) such as androgenetic alopecia (AGA) or scarring alopecia.
4. Active skin disease on the scalp or a history of skin disease on the scalp that in the opinion of the investigator would interfere with study assessments of efficacy or safety.
5. Active scalp trauma or other condition affecting the scalp that, in the investigator's opinion, may affect the course of AA, AU or AT or interfere with the study conduct or evaluations.
6. The presence of a permanent or difficult to remove hairpiece or wig that will, in the opinion of the investigator, interfere with study assessments if not removed at each visit.
7. History of, or current, severe, progressive or uncontrolled autoimmune, metabolic, hepatic, endocrine, renal, gastrointestinal, pulmonary, cardiovascular, genitourinary, or hematological disease, neurologic or cerebral disorders, or coagulation disorders that, as determined by the Investigator, would preclude participation in and completion of study assessments.
8. History of, current or suspected systemic or cutaneous malignancy and /or lymphoproliferative disease, other than subjects with a history of adequately treated and well healed and completely cleared non-melanoma skin cancers (e.g. basal or squamous cell carcinoma) treated successfully at least 1 year prior to study entry with no evidence of disease.
9. Evidence of active or latent bacterial (including tuberculosis) or viral infections at the time of enrollment, or history of incompletely treated or untreated tuberculosis. Subjects who have completed therapy for latent tuberculosis may participate.
10. History of serious local infection (e.g., cellulitis, abscess) or systemic infection including but not limited to a history of treated infection (e.g., pneumonia, septicemia) within 3 months prior to Baseline. Subjects on an antibiotic for a nonserious, acute local infection must complete the course prior to enrollment into the study.
11. Positive for HIV, Hepatitis B or C. Subjects with serologic evidence of Hepatitis B vaccination (HepB surface Ab without the presence of Hep B surface Ag will be allowed to participate).
12. History of recurrent herpes zoster (more than one episode) or disseminated herpes zoster (a single episode) or disseminated herpes simplex (single episode) or cytomegalovirus (CMV) that resolved less than 2 months before study enrollment. Subjects with a history of frequent outbreaks of Herpes Simplex Virus (defined as 4 or more outbreaks a year).
13. Subjects who have received any of the following treatments for the timeframes specified below:

    * Disease Modifying Anti-Rheumatic Drugs (DMARDS), Biologics or immunosuppressants, including but not limited to: anakinra, adalimumab, azathioprine, corticosteroids, cyclosporine, etanercept, infliximab, methotrexate, TNF inhibitors, ustekinumab within 1 month or 5 half-lives (whichever is greater) of Baseline (Visit 2).
    * Plaquenil within 2 months of Baseline (Visit 2).
    * Janus kinase (JAK) inhibitors (oral or topical) within 6 months of Baseline (Visit 2).
    * Intralesional steroids or platelet rich plasma injections in the scalp within 1 month of Baseline (Visit 2).
    * Topical treatments on the scalp with anthralin, bimatoprost, corticosteroids, diphencyprone, diphenylcyclopropenone (DPCP), squaric acid dibutylester (SADBE), minoxidil, pimecrolimus, or tacrolimus within 1 month of Baseline (Visit 2).
    * Phototherapy (narrow band Ultraviolet B [NB UVB] or broadband therapy) within 4 weeks of Baseline (Visit 2).
14. Participation in an investigational drug or device trial in which administration of an investigational drug or device occurred within 30 days or 5 half-lives (whichever is longer) of Baseline (Visit 2).
15. Any condition possibly affecting oral drug absorption, e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass. Procedures such as gastric banding are not exclusionary.
16. Unwillingness to refrain from weaves, hair extensions, or shaving of the scalp for at least two weeks prior to a study visit, at the discretion of the investigator, based on the ability to assess hair growth.
17. Vaccination with a live or attenuated vaccine within 6 weeks prior to Baseline (Visit 2) or planned vaccination with these vaccines at any time during treatment or within 6 weeks following discontinuation of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Moran, RN, Study Chair — Aclaris Therapeutics
Locations (25):
- United States (25):
  - Aclaris Investigator Site, Hot Springs, Arkansas
  - Aclaris Investigator Site, Rogers, Arkansas
  - Aclaris Investigator Site, Denver, Colorado
  - Aclaris Investigator Site, Boynton Beach, Florida
  - Aclaris Investigator Site, Miami, Florida
  - Aclaris Investigator Site, Sanford, Florida
  - Aclaris Investigator Site, Snellville, Georgia
  - Aclaris Investigator Site, Clinton Township, Michigan
  - Aclaris Investigator Site, Detroit, Michigan
  - Aclaris Investigator Site, Fridley, Minnesota
  - Aclaris Investigator Site, Minneapolis, Minnesota
  - Aclaris Investigator Site, Saint Joseph, Missouri
  - Aclaris Investigator Site, Omaha, Nebraska
  - Aclaris Investigator Site, Las Vegas, Nevada
  - Aclaris Investigator Site, New York, New York
  - Aclaris Investigator Site, Rochester, New York
  - Aclaris Investigator Site, Portland, Oregon
  - Aclaris Investigator Site, Greenville, South Carolina
  - Aclaris Investigator Site, Knoxville, Tennessee
  - Aclaris Investigator Site, Nashville, Tennessee
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigator Site, Houston, Texas
  - Aclaris Investigator Site, San Antonio, Texas
  - Aclaris Investigator Site, Lynchburg, Virginia
  - Aclaris Investigator Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-501 400mg BID Dosing: ATI-501 400mg BID dosing - oral administration
  ATI-501 400mg BID dosing: ATI-501 oral low dose
- ATI-501 600mg BID Dosing: ATI-501 600mg BID dosing - oral administration
  ATI-501 600mg BID dosing: ATI-501 oral low dose
- ATI-501 800mg BID Dosing: ATI-501 800mg BID dosing - oral administration
  ATI-501 800mg BID dosing: ATI-501 high dose for oral administration
- Placebo: Placebo: BID - oral administration
Period: Overall Study
Arm/Group | ATI-501 400mg BID Dosing | ATI-501 600mg BID Dosing | ATI-501 800mg BID Dosing | Placebo
Started | 23 | 23 | 22 | 19
Completed (Includes subjects with a SALT score after D155 occurring on or before the end of treatment date +10.) | 18 | 19 | 19 | 14
Not Completed | 5 | 4 | 3 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1
Not completed — Programmatic Analysis Non-completer | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATI-501 400mg BID Dosing | ATI-501 600mg BID Dosing | ATI-501 800mg BID Dosing | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 22 | 19 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 22 | 16 | 81
  >=65 years | 1 | 2 | 0 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.99) | 40.4 (13.56) | 40.5 (12.44) | 41.8 (16.01) | 40.3 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 13 | 14 | 56
  Male | 6 | 11 | 9 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was only sought for those subjects self-identifying as "White" when reporting their Race.
  Participants
    number analyzed (Participants) | 17 | 19 | 16 | 15 | 67
    Hispanic or Latino | 7 | 3 | 2 | 3 | 15
    Not Hispanic or Latino | 10 | 15 | 13 | 12 | 50
    Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 5 | 3 | 17
  White | 17 | 19 | 16 | 15 | 67
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 0 | 0 | 2 | 0 | 2
  II - Burns Easily | 5 | 7 | 6 | 8 | 26
  III - Burns Moderately | 7 | 9 | 4 | 8 | 28
  IV - Burns Minimally | 6 | 3 | 4 | 0 | 13
  V - Rarely Burns | 3 | 4 | 4 | 3 | 14
  VI - Never Burns | 2 | 0 | 2 | 0 | 4
Hair Pull Test - Dislodged Hairs [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 23 | 21 | 18 | 85
    Normal (≤2 hairs dislodged) | 11 | 9 | 7 | 6 | 33
    Abnormal (>2 hairs dislodged) | 0 | 5 | 1 | 1 | 7
    N/A for subjects with AU and AT (>95% hair loss) | 12 | 9 | 13 | 11 | 45
Hair pull test - broken hairs [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 23 | 21 | 18 | 85
    No | 11 | 12 | 6 | 6 | 35
    Yes | 0 | 2 | 2 | 1 | 5
    N/A for subjects with AU and AT (>95% hair loss) | 12 | 9 | 13 | 11 | 45
Hair Pull Test - Broken at Borders [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 23 | 21 | 18 | 85
    No | 11 | 12 | 6 | 6 | 35
    Yes | 0 | 2 | 2 | 1 | 5
    N/A for subjects with AU and AT (>95% hair loss) | 12 | 9 | 13 | 11 | 45
Vellus Hair Present [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 22 | 22 | 19 | 86
    No | 20 | 18 | 18 | 15 | 71
    Yes | 3 | 4 | 4 | 4 | 15
Indeterminate hair present [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 22 | 22 | 19 | 86
    No | 21 | 19 | 19 | 16 | 75
    Yes | 2 | 3 | 3 | 3 | 11
Baseline Severity of Alopecia Tool (SALT) Score Mean [Mean (Standard Deviation); unit: score on a scale] — The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth.
  score on a scale | 78 (26.7) | 76 (23.4) | 81 (25.8) | 85 (24.8) | 80 (25.0)
Baseline Severity of Alopecia Tool (SALT) Scores Percentiles [Count of Participants; unit: Participants] — The Baseline Severity of Alopecia Tool (SALT) Scores Percentiles represents the distribution of patients with SALT scores >50% (baldness affecting over half or more of the scalp) or <50% (baldness affecting less than half the scalp) at the start of the study treatment period.
  Participants
    <50% | 5 | 2 | 5 | 3 | 15
    ≥50% | 18 | 21 | 17 | 16 | 72
Baseline scalp-Patient-Reported Outcome for target patch, Alopecia Areata Patchy (AAP) subjects only [Count of Participants; unit: Participants]
  Some hair | 0 | 0 | 0 | 1 | 1
  A little hair | 8 | 8 | 5 | 4 | 25
  No hair | 3 | 6 | 4 | 3 | 16
  N/A for subjects with AU and AT (>95% hair loss) | 12 | 9 | 13 | 11 | 45
Baseline Scalp-Patient-Reported Outcome (PRO) for Entire Scalp [Count of Participants; unit: Participants]
  Most hair | 1 | 1 | 2 | 0 | 4
  Some hair | 5 | 6 | 4 | 3 | 18
  A little hair | 6 | 7 | 6 | 8 | 27
  No hair | 11 | 9 | 10 | 8 | 38
Baseline Scalp-Clinician Reported Outcomes (ClinRO) for Target Patch, AAP subjects only [Count of Participants; unit: Participants]
  A little hair | 6 | 7 | 5 | 5 | 23
  No hair | 5 | 7 | 4 | 3 | 19
  N/A for subjects with AU and AT (>95% hair loss) | 12 | 9 | 13 | 11 | 45
Baseline scalp-ClinRO for entire scalp [Count of Participants; unit: Participants]
  Some hair | 8 | 8 | 6 | 2 | 24
  A little hair | 4 | 7 | 7 | 9 | 27
  No hair | 11 | 8 | 9 | 8 | 36
Previous Therapies for Alopecia [Count of Participants; unit: Participants]
  Subjects using prior therapy for alopecia | 21 | 18 | 21 | 16 | 76
  Topical immunotherapy | 8 | 3 | 5 | 3 | 19
  Corticosteroids | 16 | 13 | 15 | 10 | 54
  Systemic steroids | 11 | 11 | 5 | 7 | 34
  DMARDS | 0 | 1 | 1 | 0 | 2
  Biologics or immunosuppressants | 0 | 1 | 0 | 1 | 2
  Plaquenil | 1 | 0 | 0 | 1 | 2
  Phototherapy | 1 | 0 | 0 | 0 | 1
  Laser therapy | 1 | 0 | 0 | 1 | 2
  NB UVB | 0 | 1 | 0 | 0 | 1
  Other | 3 | 2 | 6 | 3 | 14
Diagnosis Type [Count of Participants; unit: Participants] — AAP diagnoses were reported in the placebo group under patient Alopecia History, but only 8 of those patients had target patches identified. This discrepancy occurred due to an investigator mistakenly not collecting target patch information for a patient who was reported with a diagnosis of Alopecia Areata Patchy.
  Participants
    Alopecia Areata | 11 | 14 | 9 | 9 | 43
    Alopecia Universalis | 4 | 5 | 7 | 5 | 21
    Alopecia Totalis | 8 | 4 | 6 | 5 | 23
Ophiasis pattern of hair loss [Count of Participants; unit: Participants] — Population: The difference in the number analyzed in row differs from overall is occurring due to expected data points being omitted from collection due to site error.
  Participants
    number analyzed (Participants) | 23 | 23 | 22 | 18 | 86
    No ophiasis pattern | 19 | 19 | 18 | 17 | 73
    Ophiasis and Alopecia Areata | 4 | 4 | 4 | 1 | 13
Duration of alopecia (years) [Mean (Standard Deviation); unit: years] | 13.7 (11.01) | 9.5 (9.78) | 10.7 (11.36) | 11.3 (12.04) | 11.3 (10.94)
Duration of current episode of alopecia (weeks) [Mean (Standard Deviation); unit: weeks] | 224.2 (184.63) | 189.5 (148.31) | 176.3 (162.50) | 253.2 (153.59) | 209.3 (163.10)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair assessed by the investigator. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth by adding the percentage hair loss in the various areas (i.e. top, back, each side) of the scalp. The primary efficacy variable was the percent change from baseline in SALT score at Week 24. This was calculated as the mean of the changes from Baseline (Visit 2) SALT score to Week 24 (Visit 10) SALT score, divided by Baseline SALT score and expressed as a percentage.
Time Frame: Baseline-Week 24
Population: This primary analysis utilized the SALT score with imputation for last observation carried forward (LOCF) and was based on the intent-to-treat population.
Measure: Mean (Standard Deviation); unit: percent
Groups:
- ATI-501 400mg BID Dosing: ATI-501 400mg BID dosing (low dose) - oral administration
  ATI-501 Low dose: ATI-501 oral low dose
- ATI-501 600mg BID Dosing: ATI-501 600mg BID dosing (mid dose) - oral administration
  ATI-501 Mid dose
- ATI-501 800mg BID Dosing: ATI-501 800mg BID dosing (high dose) - oral administration
  ATI-501 high dose for oral administration
Arm/Group | ATI-501 400mg BID Dosing | ATI-501 600mg BID Dosing | ATI-501 800mg BID Dosing | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
percent | -25.6 (39.75) | -30.4 (41.23) | -25.9 (29.86) | -6.3 (23.36)
Statistical Analysis 1: Comparison: ATI-501 400mg BID Dosing vs Placebo; The planned sample size is approximately 95 enrolled subjects with approximately 45 subjects enrolled with AT or AU. Because the primary efficacy analysis of mean percent reduction in hair loss using SALT scores is expected to be more sensitive than the SALT50 responder analysis, the power for the primary analysis is also expected to be no less than 80%; Test type: Superiority; p = 0.011, Mixed Models Analysis — All statistical testing was two-sided and performed using a significance (alpha) level of 0.05; Mean Difference (Net) = -19.26, 95% CI 2-sided [-33.98 to -4.54], Standard Error of Mean 5.020
Statistical Analysis 2: Comparison: ATI-501 600mg BID Dosing vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Mixed Models Analysis — All statistical testing was two-sided and performed using a significance (alpha) level of 0.05; Mean Difference (Final Values) = -24.08, 95% CI 2-sided [-38.80 to -9.36], Standard Error of Mean 5.020
Statistical Analysis 3: Comparison: ATI-501 800mg BID Dosing vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.010, Mixed Models Analysis — All statistical testing was two-sided and performed using a significance (alpha) level of 0.05; Mean Difference (Final Values) = -19.54, 95% CI 2-sided [-34.41 to -4.67], Standard Error of Mean 5.133

2. Secondary Outcome: Percent Change From Baseline in the Alopecia Density and Extent Score (ALODEX) at Week 24
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A negative change in the ALODEX score over time represents hair regrowth.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Least Squares Mean (Standard Error); unit: percent
Groups:
- ATI-501 800mg BID Dosing: ATI-501 800mg BID Dosing (high dose) - oral administration
  ATI-501 high dose
Arm/Group | ATI-501 400mg BID Dosing | ATI-501 600mg BID Dosing | ATI-501 800mg BID Dosing | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
percent | -26.88 (5.165) | -32.24 (5.165) | -26.87 (5.281) | -7.70 (5.683)
Statistical Analysis 1: Comparison: ATI-501 400mg BID Dosing vs Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -19.17, 95% CI 2-sided [-34.33 to -4.02], Standard Error of Mean 5.165
Statistical Analysis 2: Comparison: ATI-501 600mg BID Dosing vs Placebo; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Net) = -24.53, 95% CI 2-sided [-39.69 to -9.38], Standard Error of Mean 5.165
Statistical Analysis 3: Comparison: ATI-501 800mg BID Dosing vs Placebo; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Net) = -19.17, 95% CI 2-sided [-34.48 to -3.86], Standard Error of Mean 5.281

3. Secondary Outcome: Mean Change From Baseline in the Severity of Alopecia Tool (SALT) Score at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair assessed by the investigator. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth by adding the percentage hair loss in the various areas (i.e. top, back, each side) of the scalp.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ATI-501 400mg BID: ATI-501 400mg BID Dosing (low dose) - oral administration
  ATI-501 Low dose
- ATI-501 600mg BID: ATI-501 600mg BID (mid dose) - oral administration
  ATI-501 Mid dose
- ATI-501 800mg BID: ATI-501 800mg BID (high dose) - oral administration
  ATI-501 high dose
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
score on a scale | -14.6 (23.67) | -18.6 (27.29) | -20.9 (26.50) | -3.3 (8.21)
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = -11.29, 95% CI 2-sided [-21.14 to -1.45], Standard Error of Mean 3.359
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -15.25, 95% CI 2-sided [-25.10 to -5.40], Standard Error of Mean 3.359
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -17.55, 95% CI 2-sided [-27.49 to -7.60], Standard Error of Mean 3.434

4. Secondary Outcome: Mean Change From Baseline in the Alopecia Density and Extent (ALODEX) Score at Week 24
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A negative change in the ALODEX score over time represents hair regrowth.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ATI-501 400mg BID: ATI-501 400mg BID (low dose) - oral administration
  ATI-501 Low dose
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
score on a scale | -17.6 (26.93) | -22.2 (28.99) | -20.7 (25.04) | -3.2 (8.42)
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -14.40, 95% CI 2-sided [-24.95 to -3.84], Standard Error of Mean 3.599
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -19.01, 95% CI 2-sided [-29.56 to -8.45], Standard Error of Mean 3.599
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -17.52, 95% CI 2-sided [-28.18 to -6.86], Standard Error of Mean 3.679

5. Secondary Outcome: Count of Subjects Achieving at Least a 50% Reduction in Alopecia Density and Extent (ALODEX) Score at Week 24
Description: as for outcome 4
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Vehicle - oral administration
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants | 6 | 7 | 5 | 1
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.124, Mixed Models Analysis; Odds Ratio (OR) = 4.6, 95% CI 2-sided [0.7 to 31.8]
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.079, Mixed Models Analysis; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [0.8 to 38.3]
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.177, Mixed Models Analysis; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [0.5 to 27.7]

6. Secondary Outcome: Count of Subjects in Each Treatment Arm Achieving at Least a 50% Reduction in Severity of Alopecia Tool (SALT) Score at Week 24 Compared to Baseline
Description: as for outcome 3
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants | 6 | 7 | 5 | 1
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.124, Mixed Models Analysis; Odds Ratio (OR) = 4.6, 95% CI 2-sided [0.7 to 31.8]
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.079, Mixed Models Analysis; Odds Ratio (OR) = 5.6, 95% CI 2-sided [0.8 to 38.3]
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.177, Mixed Models Analysis; Odds Ratio (OR) = 3.9, 95% CI 2-sided [0.5 to 27.7]

7. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome, Left Eyebrow
Description: The Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome is the investigator's assessment of the subject's facial hair (eyebrow(s), eyelashes,and if male, beard) at a particular point in time. The investigator was instructed to NOT refer to any other assessments to assist with these assessments. The investigator or designee assessed the affected facial hair areas (eyebrows, eyelashes and if male, beard) using a 5 point scale for each target area [1-Full (Target Area Hair); 2-Most (Target Area Hair); 3-Some (Target Area Hair); 4-A Little (Target Area Hair); 5-No (Target Area Hair)]. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 1 | 0
  Better by 3 points | 1 | 0 | 1 | 1
  Better by 2 points | 0 | 2 | 2 | 1
  Better by 1 point | 4 | 5 | 6 | 3
  No change | 15 | 15 | 10 | 13
  Worse by 1 point | 1 | 0 | 1 | 1
  Worse by 2 points | 2 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.471, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.457, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.367, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome, Right Eyebrow
Description: as for outcome 7
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebos - oral administration
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 1 | 0
  Better by 3 points | 1 | 0 | 1 | 1
  Better by 2 points | 0 | 0 | 3 | 1
  Better by 1 point | 3 | 6 | 4 | 4
  No change | 17 | 12 | 12 | 13
  Worse by 1 point | 1 | 4 | 0 | 0
  Worse by 2 points | 1 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.187, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.375, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.581, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome, Left Eyelash
Description: as for outcome 7
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Groups:
- ATI-501 600mg BID: ATI-501 600mg BID - oral administration
  ATI-501 Mid dose
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 1 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 2 | 1
  Better by 2 points | 1 | 1 | 3 | 0
  Better by 1 point | 3 | 3 | 3 | 1
  No Change | 15 | 15 | 12 | 16
  Worse by 1 point | 0 | 3 | 1 | 1
  Worse by 2 points | 1 | 0 | 0 | 0
  Worse by 3 points | 1 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.444, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.861, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.182, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome, Right Eyelash
Description: as for outcome 7
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 1 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 1 | 1
  Better by 2 points | 1 | 1 | 3 | 0
  Better by 1 point | 3 | 4 | 4 | 1
  No Change | 16 | 16 | 13 | 16
  Worse by 1 point | 0 | 1 | 0 | 1
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 1 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.258, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.263, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.101, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Clinician Reported Outcome, Beard, Male Subjects
Description: as for outcome 7
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 6 | 11 | 9 | 5
Participants
  Better by 4 points | 0 | 0 | 0 | 0
  Better by 3 points | 0 | 1 | 3 | 0
  Better by 2 points | 0 | 0 | 3 | 0
  Better by 1 point | 2 | 1 | 0 | 2
  No Change | 4 | 6 | 2 | 3
  Worse by 1 point | 0 | 2 | 1 | 0
  Worse by 2 points | 0 | 1 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.277, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.159, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome, Left Eyebrow
Description: The Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome is the patient's assessment of their facial hair (eyebrow(s), eyelashes, and if male, beard) at a particular point in time. The patient assessed the affected facial hair areas (eyebrows, eyelashes and if male, beard) using a 5 point scale for each target area [1-Full (Target Area Hair); 2-Most (Target Area Hair); 3-Some (Target Area Hair); 4-A Little (Target Area Hair); 5-No (Target Area Hair)]. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 2 | 0
  Better by 2 points | 4 | 0 | 0 | 1
  Better by 1 points | 1 | 5 | 8 | 3
  No Change | 16 | 14 | 10 | 13
  Worse by 1 point | 1 | 3 | 1 | 2
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.407, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.894, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.179, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome, Right Eyebrow
Description: as for outcome 12
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 1 | 0
  Better by 2 points | 2 | 2 | 2 | 1
  Better by 1 point | 3 | 5 | 7 | 4
  No Change | 16 | 13 | 10 | 12
  Worse by 1 point | 0 | 2 | 1 | 2
  Worse by 2 points | 1 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.691, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.521, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.262, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome, Right Eyelash
Description: as for outcome 12
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Groups:
- ATI-501 600mg BID: ATI-501 600mg BID (mid dose) - oral administration
  ATI-501 Mid dose: ATI-501 oral low dose
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 1 | 1 | 0 | 0
  Better by 3 points | 0 | 1 | 1 | 0
  Better by 2 points | 2 | 1 | 2 | 0
  Better by 1 point | 7 | 3 | 4 | 2
  No Change | 13 | 16 | 12 | 15
  Worse by 1 point | 0 | 1 | 1 | 2
  Worse by 2 points | 0 | 0 | 1 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.154, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.289, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome, Left Eyelash
Description: as for outcome 12
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 1 | 1 | 0 | 0
  Better by 3 points | 0 | 1 | 1 | 0
  Better by 2 points | 2 | 2 | 2 | 0
  Better by 1 point | 6 | 1 | 2 | 3
  No Change | 13 | 15 | 14 | 14
  Worse by 1 point | 0 | 3 | 2 | 2
  Worse by 2 points | 0 | 0 | 1 | 0
  Worse by 3 points | 1 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.073, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.660, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.704, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change From Baseline in Alopecia Facial Hair Appearance Assessment (AFHA)-Patient Reported Outcome, Beard, Male Subjects
Description: as for outcome 12
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 6 | 11 | 9 | 5
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 0 | 0 | 1 | 0
  Better by 2 points | 0 | 1 | 3 | 0
  Better by 1 point | 2 | 3 | 3 | 2
  No Change | 4 | 5 | 2 | 3
  Worse by 1 point | 0 | 1 | 0 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.911, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.110, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Change From Baseline in the Subject Global Impression of Severity (SGIS) at Week 24, Patchy Alopecia Areata
Description: The Subject Global Impression of Severity (SGIS) is a 5-point descriptive scale completed by subjects to capture the subject's assessment of disease severity at a particular timepoint. Scores of 1 to 5 are assigned to responses Mild to Extremely Severe, respectively. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 14 | 9 | 9
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 2 | 2 | 0 | 0
  Better by 2 points | 3 | 2 | 2 | 1
  Better by 1 point | 1 | 3 | 3 | 3
  No change | 3 | 5 | 3 | 4
  Worse by 1 point | 0 | 1 | 1 | 0
  Worse by 2 points | 2 | 0 | 0 | 1
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.430, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.288, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.582, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Change From Baseline in the Subject Global Impression of Severity (SGIS) at Week 24, Alopecia Universalis or Alopecia Totalis
Description: as for outcome 17
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data. One patient was excluded from the analysis based on the visit windowing conventions that was previously established. This patient's Week 24 SGIS occurred at Day 128, which is outside of the window for inclusion of results at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 9 | 13 | 10
Participants
  Better by 4 points | 0 | 1 | 1 | 0
  Better by 3 points | 1 | 0 | 3 | 0
  Better by 2 points | 2 | 1 | 2 | 0
  Better by 1 point | 2 | 0 | 3 | 2
  No change | 6 | 6 | 4 | 8
  Worse by 1 point | 0 | 1 | 0 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.194, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline in the Physician Global Impression of Severity (PhGIS) at Week 24, Patchy Alopecia Areata
Description: The Physician Global Impression of Severity (PhGIS) is a 5-point descriptive scale completed by investigators and is used to capture the investigator's assessment of the subject's disease severity at a particular timepoint. Scores of 1 to 5 are assigned to responses Mild to Extremely Severe, respectively. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 14 | 9 | 9
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 0 | 0
  Better by 2 points | 3 | 4 | 1 | 0
  Better by 1 point | 1 | 3 | 2 | 3
  No Change | 5 | 4 | 6 | 4
  Worse by 1 point | 1 | 2 | 0 | 2
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.150, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.546, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in the Physician Global Impression of Severity (PhGIS) at Week 24, Alopecia Universalis or Alopecia Totalis
Description: as for outcome 19
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 12 | 9 | 13 | 10
Participants
  Better by 4 points | 0 | 1 | 1 | 0
  Better by 3 points | 1 | 0 | 2 | 0
  Better by 2 points | 0 | 1 | 2 | 0
  Better by 1 point | 5 | 0 | 3 | 3
  No change | 6 | 7 | 5 | 7
  Worse by 1 point | 0 | 0 | 0 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.341, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.068, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Alopecia Impact Assessment (AIA) Patient Reported Outcome Change From Baseline at Week 24
Description: The Alopecia Impact Assessment (AIA) is a 13-item patient reported outcome questionnaire which measures the subject's experience with impacts related to alopecia (inclusive of all 3 subtypes observed on study) in managing appearance, worry, sadness, loss of confidence, self-consciousness, embarrassment, feeling unattractive, limitation of social activities, limitation of physical activities, unwanted attention, sweat in eyes, debris in eyes, and debris in nose. The AIA has a recall period of "over the past seven days". An 11-point NRS with anchors "0 - Not at all [impact]" and "10 - Extremely [impact]" (e.g., "Not at all bothersome" and "Extremely bothersome"; "Not at all worried" and "Extremely worried") is utilized. The AIA produces single-item (0-10) and mean total (0-10) scores, with higher scores indicating higher levels of impact.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
score on a scale | -1.9 (1.89) | -1.8 (2.79) | -1.2 (1.80) | -1.1 (1.06)

22. Secondary Outcome: Subject Global Impression of Treatment Satisfaction (SGITS) at Week 24, Patchy Alopecia Areata
Description: The Subject Global Impression of Treatment Satisfaction (SGITS) is a 7-point descriptive scale completed by subjects. Scale response options ranged from "1. Extremely Satisfied" to "7. Extremely Dissatisfied" and are used to capture how satisfied or dissatisfied they are with the study medication treatment received for their alopecia areata.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 10 | 11 | 8 | 8
Participants
  Extremely satisfied | 5 | 5 | 2 | 1
  Moderately satisfied | 2 | 2 | 2 | 0
  A little satisfied | 0 | 0 | 0 | 1
  Neither satisfied or dissatisfied | 0 | 2 | 2 | 2
  A little dissatisfied | 1 | 0 | 0 | 1
  Moderately dissatisfied | 1 | 1 | 1 | 1
  Extremely dissatisfied | 1 | 1 | 1 | 2
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.098, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.082, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.313, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Subject Global Impression of Treatment Satisfaction (SGITS) at Week 24, Alopecia Universalis or Alopecia Totalis
Description: as for outcome 22
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 12 | 9 | 13 | 10
Participants
  Extremely satisfied | 1 | 1 | 3 | 1
  Moderately satisfied | 3 | 1 | 5 | 2
  A little satisfied | 1 | 2 | 1 | 1
  Neither satisfied or dissatisfied | 4 | 3 | 1 | 3
  A little dissatisfied | 1 | 0 | 0 | 1
  Moderately dissatisfied | 1 | 1 | 1 | 1
  Extremely dissatisfied | 1 | 1 | 2 | 1
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.883, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.954, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.295, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Change From Baseline in the Subject Global Satisfaction With Hair Quality (SGSHQ) for Entire Scalp at Week 24, Patchy Alopecia Areata
Description: The investigator or study staff instructed the subject to answer the Subject Global Satisfaction with Hair Quality (SGSHQ) questionnaire in relation to their satisfaction with the quality of scalp hair at the time of questionnaire completion (ie "right now"). Subjects assessed their satisfaction with the quality of their scalp hair on a 7-point satisfaction scale from extremely satisfied to extremely dissatisfied at the visits. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 14 | 9 | 7
Participants
  Better by 6 points | 4 | 4 | 0 | 0
  Better by 5 points | 1 | 0 | 1 | 0
  Better by 4 points | 0 | 1 | 2 | 1
  Better by 3 points | 1 | 0 | 1 | 1
  Better by 2 points | 0 | 3 | 0 | 0
  Better by 1 points | 0 | 2 | 1 | 1
  No change | 4 | 4 | 2 | 4
  Worse by 1 point | 1 | 0 | 0 | 0
  Worse by 2 points | 0 | 0 | 1 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
  Worse by 5 points | 0 | 0 | 0 | 0
  Worse by 6 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.361, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.182, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.815, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Change From Baseline in the Subject Global Satisfaction With Hair Quality (SGSHQ) for Entire Scalp at Week 24, Alopecia Universalis or Alopecia Totalis
Description: as for outcome 24
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 12 | 9 | 13 | 10
Participants
  Better by 6 points | 0 | 1 | 0 | 0
  Better by 5 points | 1 | 0 | 5 | 0
  Better by 4 points | 2 | 1 | 0 | 0
  Better by 3 points | 3 | 3 | 1 | 2
  Better by 2 points | 0 | 2 | 0 | 1
  Better by 1 point | 0 | 0 | 2 | 2
  No change | 5 | 1 | 3 | 5
  Worse by 1 point | 0 | 0 | 0 | 0
  Worse by 2 points | 1 | 0 | 1 | 0
  Worse by 3 points | 0 | 0 | 1 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
  Worse by 5 points | 0 | 1 | 0 | 0
  Worse by 6 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.522, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.104, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.414, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Change in Dermatology Life Quality Index Total Score (DLQI) Between Baseline and Week 24
Description: The 10 question Dermatology Life Quality Index (DLQI) questionnaire was completed by subjects at Baseline, Week 4, Week 12, and Week 24. When completing the questionnaire, subjects were instructed to think of their hair loss in place of "skin problem" and "skin" as referenced in the questionnaire. Possible summary scores could range from 0 to 30 with higher scores indicating a worse outcome.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
score on a scale | -1.5 (4.33) | -5.3 (5.21) | -1.7 (3.97) | -1.7 (5.99)
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.882, Mixed Models Analysis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-2.53 to 2.94], Standard Error of Mean 0.930
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Net) = -3.58, 95% CI 2-sided [-6.31 to -0.84], Standard Error of Mean 0.930
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.999, Mixed Models Analysis; Mean Difference (Net) = 0.00, 95% CI 2-sided [-2.76 to 2.76], Standard Error of Mean 0.951

27. Secondary Outcome: Subject Global Impression of Change (SGIC) at Week 24
Description: The Subject Global Impression of Change (SGIC) is a 7-point descriptive scale completed by subjects at Week 24 (Intent-to-treat population with reported data falling within the windowed Week 24 visit timeframe). Scale response options ranged from "1. Very much improved" to "7. Very much worse" and are used to capture the subject's overall impression of change for his/her alopecia during the treatment period.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward (LOCF) to address missing data. Per SAP, the allowed window days for Week 24 visit are 155-182. There were 4 patients in the 400mg group, 4 patients in the 600mg group, 3 patients in the 800mg group, and 5 patients in the placebo group who fell outside this window.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 14
Participants
  Very much improved | 5 | 6 | 2 | 1
  Much improved | 3 | 1 | 7 | 1
  A little improved | 4 | 5 | 6 | 6
  No change | 7 | 7 | 3 | 6
  A little worse | 0 | 0 | 1 | 0
  Much worse | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.270, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.319, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.094, Wilcoxon (Mann-Whitney)

28. Secondary Outcome: Physician Global Impression of Change (PhGIC) at Week 24
Description: The Physician Global Impression of Change (PhGIC) is a 7-point descriptive scale completed by investigators at Week 24 (Intent-to-treat population with reported data falling within the windowed Week 24 visit timeframe). Scale response options ranged from "1. Very much improved" to "7. Very much worse" and are used to capture the investigator's overall impression of change for the subject's alopecia during the treatment period.
Time Frame: Baseline-Week 24
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 14
Participants
  Very much improved | 5 | 7 | 3 | 2
  Much improved | 3 | 0 | 6 | 0
  A little improved | 2 | 5 | 5 | 5
  No change | 8 | 7 | 4 | 7
  A little worse | 1 | 0 | 1 | 0
  Much worse | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.584, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.287, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.144, Wilcoxon (Mann-Whitney)

29. Secondary Outcome: Change From Baseline in Alopecia Scalp Appearance Assessment (ASAA): Scalp-Clinician Reported Outcome for Target Patch, Patchy Alopecia Areata
Description: The Scalp Clinician Reported Outcome for Target Patch provides the investigator's assessment for Patchy Alopecia Areata (AAP) patients regarding the appearance of the patient's target patch (identified by the patient as his or her most bothersome area of scalp hair loss at Baseline). The assessment was completed by investigators at Baseline, Week 2, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, scalp of the target patch completely covered with hair" to "no hair, scalp of the target patch completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the patient's target patch. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 14 | 9 | 8
Participants
  Better by 4 points | 0 | 1 | 1 | 0
  Better by 3 points | 4 | 5 | 1 | 2
  Better by 2 points | 1 | 1 | 0 | 0
  Better by 1 point | 0 | 3 | 4 | 0
  No change | 6 | 2 | 2 | 5
  Worse by 1 point | 0 | 2 | 1 | 1
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.341, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.203, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.327, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline in Alopecia Scalp Appearance Assessment (ASAA): Scalp-Clinician Reported Outcome for Entire Scalp, All Patients
Description: The Scalp Clinician Reported Outcome for Entire Scalp was completed for patients with Patchy Alopecia Areata, Alopecia Universalis, and Alopecia Totalis and assesses the appearance of the patient's whole scalp. The assessment was completed by investigators at Baseline, Week 2, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, whole scalp completely covered with hair" to "no hair, whole scalp completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the patient's whole scalp. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 1 | 0 | 1 | 0
  Better by 2 points | 3 | 2 | 3 | 1
  Better by 1 point | 7 | 9 | 8 | 8
  No change | 11 | 10 | 10 | 10
  Worse by 1 point | 1 | 1 | 0 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.827, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.742, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.462, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Change From Baseline in Alopecia Scalp Appearance Assessment (ASAA): Scalp-Patient Reported Outcome for Target Patch, Patchy Alopecia Areata
Description: The Scalp Patient Reported Outcome for Target Patch was completed by patients with Patchy Alopecia Areata (AAP) and assesses the appearance of the subject's target patch (identified by the subject as his or her most bothersome area of scalp hair loss at Baseline). The assessment was completed by AAP subjects at Baseline, Week 2, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, scalp of the target patch completely covered with hair" to "no hair, scalp of the target patch completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the subject's target patch. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 11 | 14 | 9 | 8
Participants
  Better by 4 points | 2 | 1 | 1 | 0
  Better by 3 points | 3 | 4 | 1 | 1
  Better by 2 points | 1 | 3 | 0 | 1
  Better by 1 point | 0 | 2 | 4 | 5
  No change | 4 | 1 | 2 | 1
  Worse by 1 point | 1 | 3 | 1 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.836, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.540, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.672, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: Change From Baseline in Alopecia Scalp Appearance Assessment (ASAA): Scalp-Patient Reported Outcome for Entire Scalp, All Patients
Description: The Scalp Patient Reported Outcome for Entire Scalp was completed by patients with Patchy Alopecia Areata, Alopecia Universalis, and Alopecia Totalis and assesses the appearance of the patient's whole scalp. The assessment was completed by patients at Baseline, Week 2, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, whole scalp completely covered with hair" to "no hair, whole scalp completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the patient's target patch. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline-Week 24
Population: Intent-to-treat population using Last Observation Carried Forward to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-501 400mg BID | ATI-501 600mg BID | ATI-501 800mg BID | Placebo
Number analyzed (Participants) | 23 | 23 | 22 | 19
Participants
  Better by 4 points | 0 | 1 | 0 | 0
  Better by 3 points | 2 | 1 | 1 | 0
  Better by 2 points | 4 | 2 | 5 | 1
  Better by 1 point | 5 | 10 | 7 | 7
  No change | 11 | 8 | 8 | 11
  Worse by 1 point | 1 | 1 | 1 | 0
  Worse by 2 points | 0 | 0 | 0 | 0
  Worse by 3 points | 0 | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: ATI-501 400mg BID vs Placebo; Test type: Superiority; p = 0.469, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ATI-501 600mg BID vs Placebo; Test type: Superiority; p = 0.219, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ATI-501 800mg BID vs Placebo; Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Double blind period = 24 weeks; Reporting of non-serious AEs started with each subject's first study medication application and continued until the 30 days after the subject's last study visit. Reporting for SAEs started when the subject signed the informed consent document and continued until 30 days after the subject's last visit.
Arm/Group | ATI-501 400mg BID Dosing | ATI-501 600mg BID Dosing | ATI-501 800mg BID Dosing | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 5/23 | 2/23 | 3/22 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-501 400mg BID Dosing (N=23) | ATI-501 600mg BID Dosing (N=23) | ATI-501 800mg BID Dosing (N=22) | Placebo (N=19)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03594227/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03594227/SAP_001.pdf
  • Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03594227/ICF_002.pdf